CLINICAL TRIAL: NCT01657461
Title: Solitaire™ FR With the Intention For Thrombectomy as Primary Endovascular Treatment for Acute Ischemic Stroke (SWIFT PRIME) Clinical Trial
Brief Title: Solitaire™ With the Intention For Thrombectomy as PRIMary Endovascular Treatment (SWIFT PRIME) Trial
Acronym: SWIFT PRIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV-SFR004
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-04

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV t-PA with Solitaire™ revascularization device (Experimental): Dual IV tPA therapy and adjunctive treatment with the Solitaire revascularization device
  Interventions: Device: Solitaire revascularization device
- IV t-PA (Active Comparator): Infusion of intravenous tissue plasminogen activator (IV t-PA)
  Interventions: Drug: Intravenous (IV) recombinant human tissue plasminogen activator (rtPA)

INTERVENTIONS:
Drug: Intravenous (IV) recombinant human tissue plasminogen activator (rtPA) — Standard therapy with Intravenous (IV) recombinant human tissue plasminogen activator (rtPA)
  Arms: IV t-PA
Device: Solitaire revascularization device — Clot retrieval with the Solitaire revascularization device after patients have received standard therapy with intravenous tissue plasminogen activator
  Arms: IV t-PA with Solitaire™ revascularization device

SUMMARY:
The primary study objective is to determine if subjects experiencing an acute ischemic stroke due to large vessel occlusion, treated with combined IV t-PA and Solitaire Revascularization Device within 6 hours of symptom onset have less stroke-related neurological disability (mRS) than those subjects treated with IV t-PA alone

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 80
2. Clinical signs consistent with acute ischemic stroke
3. Prestroke Modified Rankin Score ≤ 1
4. NIHSS ≥ 8 and < 30 at the time of randomization
5. Initiation of IV t-PA within 4.5 hours of onset of stroke symptoms (onset time is defined as the last time when the patient was witnessed to be at baseline), with investigator verification that the subject has received / is receiving the correct IV t-PA dose for the estimated weight prior to randomization.
6. Thrombolysis in Cerebral Infarction (TICI) 0-1 flow in the intracranial internal carotid artery, M1 segment of the MCA, or carotid terminus confirmed by CT or MR angiography that is accessible to the Solitaire™ FR Device.
7. Subject is able to be treated within 6 hours of onset of stroke symptoms and within 1.5 hours (90 minutes) from CTA or MRA to groin puncture.
8. Subject is willing to conduct protocol-required follow-up visits.
9. An appropriate signed and dated Informed Consent Form (as allowed according to country regulations and approved by ethics committee and/or IRB) has been obtained
10. Subject is affiliated with a social security system (if required by individual country regulations).
11. Subject meets national regulatory criteria for clinical trial participation.

Exclusion Criteria:

1. Subject who is contraindicated to IV t-PA as per local national guidelines.
2. Female who is pregnant or lactating or has a positive pregnancy test at time of admission.
3. As applicable by French law, subject who is a protected individual such as an incompetent adult or incarcerated person.
4. Rapid neurological improvement prior to study randomization suggesting resolution of signs/symptoms of stroke.
5. Known serious sensitivity to radiographic contrast agents.
6. Known sensitivity to Nickel, Titanium metals or their alloys.
7. Current participation in another investigational drug or device treatment study.
8. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency. (A subject without history or suspicion of coagulopathy does not require INR or prothrombin time lab results to be available prior to enrollment.)
9. Renal Failure as defined by a serum creatinine > 2.0 mg/dl (or 176.8 μmol/l) or Glomerular Filtration Rate [GFR] < 30Warfarin therapy with INR greater than 1.7.
10. Subject who requires hemodialysis or peritoneal dialysis, or who have a contraindication to an angiogram for whatever reason
11. Life expectancy of less than 90 days.
12. Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT or MRI scan is normal.
13. Suspicion of aortic dissection.
14. Subject with a co-morbid disease or condition that would confound the neurological and functional evaluations or compromise survival or ability to complete follow-up assessments.
15. Subject currently uses or has a recent history of illicit drug(s) or abuses alcohol (defined as regular or daily consumption of more than 4 alcoholic drinks per day).
16. Known history of arterial tortuosity, pre-existing stent, and/or other arterial disease which would prevent the device from reaching the target vessel and/or preclude safe recovery of the device.

Imaging Exclusion Criteria:

1. Computed tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of hemorrhage on presentation.
2. CT or MRI evidence of mass effect or intra-cranial tumor (except small meningioma).
3. CT or MRI evidence of cerebral vasculitis.
4. CT showing hypodensity or MRI showing hyperintensity involving greater than 1/3 of the middle cerebral artery (MCA) territory (or in other territories, >100 cc of tissue) on presentation.
5. Baseline non-contrast CT or DWI MRI evidence of a moderate/large core defined as extensive early ischemic changes of Alberta Stroke Program Early CT score (ASPECTS) < 6.
6. CT or MRI evidence of a basilar artery (BA) occlusion or posterior cerebral artery (PCA) occlusion.
7. CTA or MRA evidence of carotid dissection or complete cervical carotid occlusion requiring stenting at the time of the index procedure (i.e., mechanical thrombectomy)
8. Imaging evidence that suggests, in the opinion of the investigator, the subject is not appropriate for mechanical thrombectomy intervention (e.g., inability to navigate to target lesion, moderate/large infarct with poor collateral circulation, etc).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2012-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Saver, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Kaleida Health/Buffalo General, Buffalo, New York, United States

REFERENCES:
- [Derived] Raychev R, Saver JL, Jahan R, Nogueira RG, Goyal M, Pereira VM, Gralla J, Levy EI, Yavagal DR, Cognard C, Liebeskind DS. The impact of general anesthesia, baseline ASPECTS, time to treatment, and IV tPA on intracranial hemorrhage after neurothrombectomy: pooled analysis of the SWIFT PRIME, SWIFT, and STAR trials. J Neurointerv Surg. 2020 Jan;12(1):2-6. doi: 10.1136/neurintsurg-2019-014898. Epub 2019 Jun 25. PMID 31239326
- [Derived] Eker OF, Saver JL, Goyal M, Jahan R, Levy EI, Nogueira RG, Yavagal DR, Bonafe A; SWIFT PRIME investigators. Impact of Anesthetic Management on Safety and Outcomes Following Mechanical Thrombectomy for Ischemic Stroke in SWIFT PRIME Cohort. Front Neurol. 2018 Aug 29;9:702. doi: 10.3389/fneur.2018.00702. eCollection 2018. PMID 30210431
- [Derived] Kaneko N, Komuro Y, Yokota H, Tateshima S. Stent retrievers with segmented design improve the efficacy of thrombectomy in tortuous vessels. J Neurointerv Surg. 2019 Feb;11(2):119-122. doi: 10.1136/neurintsurg-2018-014061. Epub 2018 Jul 24. PMID 30045949
- [Derived] Arenillas JF, Cortijo E, Garcia-Bermejo P, Levy EI, Jahan R, Liebeskind D, Goyal M, Saver JL, Albers GW. Relative cerebral blood volume is associated with collateral status and infarct growth in stroke patients in SWIFT PRIME. J Cereb Blood Flow Metab. 2018 Oct;38(10):1839-1847. doi: 10.1177/0271678X17740293. Epub 2017 Nov 14. PMID 29135347
- [Derived] Raychev R, Jahan R, Saver JL, Nogueira RG, Goyal M, Pereira VM, Levy E, Yavagal DR, Cognard C, Liebeskind D. Microcatheter contrast injection in stent retriever neurothrombectomy is safe and useful: insights from SWIFT PRIME. J Neurointerv Surg. 2018 Jul;10(7):615-619. doi: 10.1136/neurintsurg-2017-013397. Epub 2017 Nov 10. PMID 29127195
- [Derived] Menjot de Champfleur N, Saver JL, Goyal M, Jahan R, Diener HC, Bonafe A, Levy EI, Pereira VM, Cognard C, Yavagal DR, Albers GW. Efficacy of Stent-Retriever Thrombectomy in Magnetic Resonance Imaging Versus Computed Tomographic Perfusion-Selected Patients in SWIFT PRIME Trial (Solitaire FR With the Intention for Thrombectomy as Primary Endovascular Treatment for Acute Ischemic Stroke). Stroke. 2017 Jun;48(6):1560-1566. doi: 10.1161/STROKEAHA.117.016669. Epub 2017 May 2. PMID 28465460
- [Derived] Mokin M, Levy EI, Saver JL, Siddiqui AH, Goyal M, Bonafe A, Cognard C, Jahan R, Albers GW; SWIFT PRIME Investigators. Predictive Value of RAPID Assessed Perfusion Thresholds on Final Infarct Volume in SWIFT PRIME (Solitaire With the Intention for Thrombectomy as Primary Endovascular Treatment). Stroke. 2017 Apr;48(4):932-938. doi: 10.1161/STROKEAHA.116.015472. Epub 2017 Mar 10. PMID 28283606
- [Derived] Shireman TI, Wang K, Saver JL, Goyal M, Bonafe A, Diener HC, Levy EI, Pereira VM, Albers GW, Cognard C, Hacke W, Jansen O, Jovin TG, Mattle HP, Nogueira RG, Siddiqui AH, Yavagal DR, Devlin TG, Lopes DK, Reddy VK, du Mesnil de Rochemont R, Jahan R, Vilain KA, House J, Lee JM, Cohen DJ; SWIFT-PRIME Investigators. Cost-Effectiveness of Solitaire Stent Retriever Thrombectomy for Acute Ischemic Stroke: Results From the SWIFT-PRIME Trial (Solitaire With the Intention for Thrombectomy as Primary Endovascular Treatment for Acute Ischemic Stroke). Stroke. 2017 Feb;48(2):379-387. doi: 10.1161/STROKEAHA.116.014735. Epub 2016 Dec 27. PMID 28028150
- [Derived] Albers GW, Goyal M, Jahan R, Bonafe A, Diener HC, Levy EI, Pereira VM, Cognard C, Yavagal DR, Saver JL. Relationships Between Imaging Assessments and Outcomes in Solitaire With the Intention for Thrombectomy as Primary Endovascular Treatment for Acute Ischemic Stroke. Stroke. 2015 Oct;46(10):2786-94. doi: 10.1161/STROKEAHA.115.010710. Epub 2015 Aug 27. PMID 26316344
- [Derived] Saver JL, Goyal M, Bonafe A, Diener HC, Levy EI, Pereira VM, Albers GW, Cognard C, Cohen DJ, Hacke W, Jansen O, Jovin TG, Mattle HP, Nogueira RG, Siddiqui AH, Yavagal DR, Baxter BW, Devlin TG, Lopes DK, Reddy VK, du Mesnil de Rochemont R, Singer OC, Jahan R; SWIFT PRIME Investigators. Stent-retriever thrombectomy after intravenous t-PA vs. t-PA alone in stroke. N Engl J Med. 2015 Jun 11;372(24):2285-95. doi: 10.1056/NEJMoa1415061. Epub 2015 Apr 17. PMID 25882376

RESULTS

PARTICIPANT FLOW:
Groups:
- IV t-PA With Solitaire™ Revascularization Device: Dual IV tPA therapy and adjunctive treatment with the Solitaire™ FR
- IV t-PA: IV infusion of tPA
Period: Overall Study
Arm/Group | IV t-PA With Solitaire™ Revascularization Device | IV t-PA
Started | 98 | 98
Completed | 88 | 78
Not Completed | 10 | 20
Not completed — Death | 9 | 12
Not completed — Lost to Follow-up | 0 | 3
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: Two subjects in the IV t-PA arm withdrew and requested all data removed and was not included in analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | IV t-PA With Solitaire™ Revascularization Device | IV t-PA | Total
Number analyzed (Participants) | 98 | 96 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Date of birth was not recorded per country regulations.
  years
    number analyzed (Participants) | 98 | 95 | 193
    (all) | 64.99 (12.49) | 66.32 (11.277) | 65.64 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 51 | 95
  Male | 54 | 45 | 99
Region of Enrollment [Number; unit: participants]
  United States | 65 | 66 | 131
  Austria | 1 | 1 | 2
  Denmark | 1 | 1 | 2
  France | 8 | 4 | 12
  Germany | 20 | 22 | 42
  Spain | 1 | 1 | 2
  Switzerland | 2 | 1 | 3
NIHSS [Mean (Standard Deviation); unit: Scores on a scale] — The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. NIHSS scores range from 0 - 42. A score of 0 indicates no stroke symptoms. Higher scores indicate incremental levels of neurological impairment. Population: Two subjects in the IV t-PA arm did not have baseline NIHSS recorded
  Scores on a scale
    number analyzed (Participants) | 98 | 94 | 192
    (all) | 16.69 (4.68) | 16.49 (4.60) | 16.59 (4.63)

OUTCOME MEASURES:

1. Primary Outcome: 90-day Global Disability Assessed Via the Blinded Evaluation of Modified Rankin Score (mRS).
Description: mRS is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke. 0 No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Time Frame: 90 days
Population: Final assessment unavailable for 5 subjects that withdrew consent or investigator withdrew consent in IV t-PA arm.
Measure: Count of Participants; unit: Participants
Arm/Group | IV t-PA With Solitaire™ Revascularization Device | IV t-PA
Number analyzed (Participants) | 98 | 93
Participants
  mRS 0 | 17 | 8
  mRS 1 | 25 | 10
  mRS 2 | 17 | 15
  mRS 3 | 12 | 16
  mRS 4 | 15 | 20
  mRS 5/6 | 12 | 24

2. Secondary Outcome: Death Due to Any Cause at 90 Days
Time Frame: 90 days
Population: One subject in the IV t-PA arm withdrew and requested all data be removed.
Measure: Count of Participants; unit: Participants
Arm/Group | IV t-PA With Solitaire™ Revascularization Device | IV t-PA
Number analyzed (Participants) | 98 | 97
Participants | 9 | 12

3. Secondary Outcome: Functional Independence as Defined by Modified Rankin Scale (mRS) Score ≤2 at 90 Days
Time Frame: 90 days
Population: Final assessment unavailable for 5 subjects that withdrew consent or investigator withdrew consent in IV t-PA arm.
Measure: Count of Participants; unit: Participants
Arm/Group | IV t-PA With Solitaire™ Revascularization Device | IV t-PA
Number analyzed (Participants) | 98 | 93
Participants | 59 | 33

4. Secondary Outcome: Change in NIH Stroke Scale Score at 27 ± 6 Hrs Post Randomization
Description: The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. NIHSS scores range from 0 - 42. A score of 0 indicates no stroke symptoms. Higher scores indicate incremental levels of neurological impairment.
Time Frame: Baseline to 27±6 hours post randomization
Population: Final assessment not available for all subjects.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IV t-PA With Solitaire™ Revascularization Device | IV t-PA
Number analyzed (Participants) | 97 | 92
units on a scale | -8.5 (7.1) | -3.9 (6.2)

5. Secondary Outcome: Volume of Cerebral Infarction as Measured by a CT or MRI Scan at 27±6 Hours Post Randomization
Time Frame: 27±6 hours post randomization
Population: Final assessment not available for all subjects.
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | IV t-PA With Solitaire™ Revascularization Device | IV t-PA
Number analyzed (Participants) | 97 | 94
cc | 60.2 (86) | 65.9 (73.5)

6. Secondary Outcome: Reperfusion Measured by Reperfusion Ratio on CT or MRI Scan 27±6 Hours Post Randomization
Time Frame: 27±6 hours post randomization
Population: Final assessment not available for all subjects.
Measure: Mean (Standard Deviation); unit: Reperfusion ratio
Arm/Group | IV t-PA With Solitaire™ Revascularization Device | IV t-PA
Number analyzed (Participants) | 64 | 52
Reperfusion ratio | 81 (67.3) | 61.9 (53)

7. Secondary Outcome: Arterial Revascularization Measured by TICI 2b or 3 Following Device Use
Time Frame: Post procedure
Population: Final assessment not available for all subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | IV t-PA With Solitaire™ Revascularization Device | IV t-PA
Number analyzed (Participants) | 83 | 0
Participants | 73 |

8. Secondary Outcome: Correlation of RAPID-assessed Core Infarct Volume With 27±6 Hours Post Randomization Stroke Infarction in Subjects Who Achieved TICI 2b-3 Reperfusion Without Intracranial Hemorrhage
Time Frame: 27±6 hours post randomization
Population: Final assessment not available for all subjects.
Measure: Number; unit: Correlation
Arm/Group | IV t-PA With Solitaire™ Revascularization Device | IV t-PA
Number analyzed (Participants) | 58 | 0
Correlation | 0.46 |

9. Other Pre Specified Outcome: Incidence of All Serious Adverse Events (SAEs)
Time Frame: Through 90 days
Population: One subject in the IV t-PA arm withdrew and requested all data be removed.
Measure: Count of Participants; unit: Participants
Arm/Group | IV t-PA With Solitaire™ Revascularization Device | IV t-PA
Number analyzed (Participants) | 98 | 97
Participants | 35 | 30

10. Other Pre Specified Outcome: Incidence of sICH at 27±6 Hours Post Randomization
Time Frame: 27±6 hours post randomization
Population: One subject in the IV t-PA arm withdrew and requested all data be removed.
Measure: Count of Participants; unit: Participants
Arm/Group | IV t-PA With Solitaire™ Revascularization Device | IV t-PA
Number analyzed (Participants) | 98 | 97
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | IV t-PA With Solitaire™ Revascularization Device | IV t-PA
Serious Adverse Events (participants affected / at risk) | 35/98 | 30/97
Other Adverse Events (participants affected / at risk) | 91/98 | 88/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV t-PA With Solitaire™ Revascularization Device (N=98) | IV t-PA (N=97)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 2 (2) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 2 (2) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 3 (3) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 4 (4)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (3) | 6 (6)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Stroke in evolution (Nervous system disorders) | 7 (7) | 8 (8)
Vasculitis cerebral (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 2 (2)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Arterial rupture (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery embolism (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vascular occlusion (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV t-PA With Solitaire™ Revascularization Device (N=98) | IV t-PA (N=97)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 4 (4)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 6 (6) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 5 (5)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 4 (4) | 7 (8)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 2 (2) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 8 (8) | 9 (9)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Optic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 17 (18) | 15 (16)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 8 (8) | 8 (8)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (9) | 6 (6)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (7) | 4 (4)
Application site pruritus (General disorders) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Catheter site induration (General disorders) | 1 (1) | 0 (0)
Catheter site inflammation (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0)
Extravasation (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (4) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Local swelling (General disorders) | 2 (2) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 4 (4)
Pain (General disorders) | 5 (5) | 3 (3)
Polyp (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 9 (9) | 7 (7)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (1)
Temperature intolerance (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 2 (2)
Immune system disorder (Immune system disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridium colitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 2 (2) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 3 (3) | 4 (4)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 13 (14) | 8 (8)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 3 (3)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 19 (21) | 29 (33)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 3 (3)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tracheal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Biopsy salivary gland (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood magnesium abnormal (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 9 (10) | 8 (8)
Blood urea increased (Investigations) | 1 (1) | 1 (1)
Cardiac enzymes increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ST segment abnormal (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 2 (2) | 2 (2)
Troponin increased (Investigations) | 2 (2) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 4 (4) | 7 (7)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 18 (18) | 7 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 3 (3) | 2 (2)
Carotid artery dissection (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral vasoconstriction (Nervous system disorders) | 12 (12) | 0 (0)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 2 (2)
Convulsion (Nervous system disorders) | 1 (1) | 6 (6)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 32 (33) | 39 (40)
Headache (Nervous system disorders) | 16 (17) | 16 (16)
Hemianopia (Nervous system disorders) | 1 (1) | 1 (1)
Horner's syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Hypertonia (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 2 (2) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 2 (2) | 2 (2)
Intraventricular haemorrhage (Nervous system disorders) | 4 (4) | 3 (3)
Ischaemic stroke (Nervous system disorders) | 3 (4) | 9 (9)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1)
Muscle spasticity (Nervous system disorders) | 2 (2) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Stroke in evolution (Nervous system disorders) | 8 (8) | 8 (8)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Vasculitis cerebral (Nervous system disorders) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 6 (6) | 8 (8)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (3) | 4 (4)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 15 (15) | 15 (15)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 9 (9) | 5 (5)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 3 (3)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 5 (5) | 4 (4)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 9 (9) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Gastrostomy tube removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Arterial rupture (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 8 (8) | 7 (7)
Embolism arterial (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery embolism (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 4 (4)
Hypotension (Vascular disorders) | 6 (6) | 6 (6)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 3 (3) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vascular occlusion (Vascular disorders) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Physician shall not make any publication without providing Sponsor 30 days notice.If Sponsor determines that the proposed publication contains confidential information, Sponsor may require the delay of publication for a period of time not to exceed 90 days and may require that any confidential information be removed from the publication. Sponsor may also require Physician to delay publication until any factual errors or inaccuracies in the publication are corrected.